CLINICAL TRIAL: NCT01099462
Title: Ibuprofen Concentration in Cerebro Spinal Fluid (CSF) of Infants and Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Eran Kozer, Assaf harofeh Medical center
Other Study IDs: 199/07*3
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-03

CONDITIONS: Fever
Keywords: fever; Ibuprofen
MeSH Terms: conditions — Fever | interventions — Ibuprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood CSF
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with fever
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen (10mg/kg BW) will be given orally if the temperature on presentation is higher than 38.0OC according to the decision of the attending physician.

SUMMARY:
Ibuprofen, the active ingredient in Nurofen and Advil, is a commonly used drug in children. There is very limited data about Ibuprofen concentrations in the cerebro spinal fluid (CSF). The objective of the current study is to describe concentrations of ibuprofen in the CSF of infants and children after administration of ibuprofen. We will study infants presenting to the Emergency Department (ED) with fever who received ibuprofen. A complete sepsis workup including sampling of blood and CSF is conducted in cases of suspected meningitis. We will measure ibuprofen in the blood and CSF obtained during the sepsis workup. A better understanding of the pharmacokinetics of ibuprofen and its penetration into the CSF will unable us to suggest more accurate dosing guidelines, and to better predict the effects of this commonly used drug.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3 month-18 years
* Rectal temperature > 38.0OC or oral temperature > 37.6 OC measured in the ED or at home.
* A sepsis work up is indicated
* At least one dose of Ibuprofen was given in the last 8 hours prior to lumbar puncture (LP)

Exclusion Criteria:

* Hypersensitivity to Ibuprofen
* Known metabolic disorder
* Known liver or kidney disease
* Hydrocephalus
* Informed consent could not be obtained from a legal guardian

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and Infants 3 month to 18 years of age with fever (rectal temperature >38.0OC or oral temperature > 37.6 OC)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Ibuprofen concentration in the CSF | 30 - 360 minutes after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh, Ẕerifin, Israel

REFERENCES:
- [Derived] Har-Even R, Stepensky D, Britzi M, Soback S, Chaim AB, Brandriss N, Goldman M, Berkovitch M, Kozer E. Plasma and cerebrospinal fluid concentrations of ibuprofen in pediatric patients and antipyretic effect: Pharmacokinetic-pharmacodynamic modeling analysis. J Clin Pharmacol. 2014 Sep;54(9):1023-30. doi: 10.1002/jcph.307. Epub 2014 Apr 21. PMID 24733245